CLINICAL TRIAL: NCT01570361
Title: Atrial Fibrillation Progression Trial
Acronym: ATTEST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The sponsor decided to terminate the study early due to enrolment not proceeding in accordance with expectations, independently from the study outcome.
Sponsor: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATTEST
Record Dates: First submitted 2012-03-28; First posted 2012-04-04 (Estimated); Results first posted 2020-05-14 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Pathologic Processes
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases; Pathologic Processes | interventions — Catheter Ablation; Anti-Arrhythmia Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Catheter Ablation (Experimental): Radiofrequency catheter ablation treatment in subjects with Paroxysmal Atrial Fibrillation (PAF)
  Interventions: Device: Catheter Ablation
- Drug Treatment (Active Comparator): Drug therapy (either rate or rhythm control) using current AF management guidelines
  Interventions: Drug: Drug Treatment

INTERVENTIONS:
Device: Catheter Ablation — Treat subjects with Paroxysmal Atrial Fibrillation (PAF)
  Other Names: CARTO® 3 or CARTO® XP System and THERMOCOOL® Catheter Family
  Arms: Catheter Ablation
Drug: Drug Treatment — Drug therapy (either rate or rhythm control): Class I or class III, or AV nodal blocking agents such as beta blockers and calcium channel blockers in accordance with current atrial fibrillation management guidelines.
  Other Names: Antiarrhythmic Drugs
  Arms: Drug Treatment

SUMMARY:
The objective of this study is to determine whether early radiofrequency (RF) ablation treatment, using the CARTO® 3 or CARTO® XP System, and THERMOCOOL® Catheter Family (including THERMOCOOL® SF or THERMOCOOL® SMARTTOUCH™) in subjects with paroxysmal atrial fibrillation (PAF), delays progression of atrial fibrillation (AF) compared with drug therapy (either rate or rhythm control) using current AF management guidelines.

DETAILED DESCRIPTION:
Eligible PAF subjects with recurrent AF for 2 years who have failed no more than 2 prescribed drugs (with either anti-arrhythmic or rate control drug) are randomized into one of two study arms (catheter ablation or drug therapy).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent paroxysmal atrial fibrillation (AF) for at least 2 years, with ≥ 2 episodes over the last 6 months; (per Amendment v3, 09APR2013, previous "6 episodes" )
2. HATCH Score of at least ≥1 and ≤4.
3. Eligible for catheter ablation and for anti-arrhythmic or rate control medications, after having failed at least 1 but no more than 2 prescribed drugs (either anti-arrhythmic or rate control drug).
4. Age 60 years or older.
5. Left atrium (LA) diameter ≤ 55mm by TTE.
6. Left ventricle (LV) ejection fraction ≥50% when in sinus rhythm or LV ejection fraction ≥35% when in atrial fibrillation.

   NOTE: For patients entering the study in AF with an ejection fraction ≥35% and <50%; the ejection fraction should be re-checked when in sinus rhythm. In case the ejection fraction is >50% the subject can continue in the study.
7. Patient signed the Informed Consent Form and is able and willing to comply with protocol requirements, including all baseline and follow-up testing.

Exclusion Criteria:

1. Patients awaiting cardiac transplantation or other cardiac surgery.
2. Acute illness (ongoing) or active systemic infection or sepsis which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant of the study.
3. Reversible causes of atrial fibrillation, e.g. but not limited to thyroid disorders, acute alcohol intoxication, recent major surgical procedures or trauma, etc.
4. Recent cardiac events including myocardial infarction (MI), percutaneous coronary intervention (PCI), or valve or bypass surgery in the preceding 3 months.
5. Heart failure decompensation.
6. Previously diagnosed with persistent/permanent atrial fibrillation/ atrial flutter.
7. Previously required cardioversion >48 hours after onset of atrial fibrillation/ atrial flutter.
8. Subject having previous transischemic attack (TIA) or stroke (cerebrovascular accident) one year prior to patient enrolment and/or no sufficient recovery.
9. Pulmonary embolism or recent atrial embolism/thrombosis.
10. Hypertrophic obstructive cardiomyopathy.
11. Class IV angina or Class IV congestive heart failure (CHF) (including past or planned heart transplantation).
12. Mandated anti-arrhythmic drug therapy for disease conditions other than atrial fibrillation.
13. Heritable arrhythmias or increased risk for torsade de pointes with class I or III Drugs.
14. Prior left atrial catheter ablation with the intention of treating atrial fibrillation; prior surgical interventions for AF such as the MAZE procedure.
15. Prior AV nodal ablation.
16. Patients presenting contra-indications for the study catheter(s), as indicated in the respective Instructions For Use.
17. Contraindication to warfarin, other anticoagulation therapy, or all anti-platelet medications.
18. Medical conditions limiting expected survival to <3 years.
19. Concurrent participation in any other clinical study.
20. Prior history of non-adherence to prescribed drug regimens.
21. Women of child bearing potential whom are pregnant, lactating, or planning to become pregnant during the course of the trial

NOTE: Prior ablation of the cavo-tricuspid isthmus is not a reason to exclude, if the patient develops subsequent recurrent atrial fibrillation.

NOTE: For patients randomized to the PVI group (Test Group), a Transesophageal Echocardiography (TEE) should be performed (as per standard of care), within 48 hours pre-procedure, to exclude atrial thrombus or other structural contraindications for an ablation procedure.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2012-02-13 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Kuck, MD, Principal Investigator — Asklepios Klinik St. Georg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled on 13-Feb-2012. On 27-Feb-2018, study was terminated early due to enrollment not proceeding in accordance with expectations, independently from the study outcome. The last subject completed the last visit on 29-May-2018.
Pre-assignment Details: Before randomization and signing inform consent forms, all subjects were screened according protocol defined inclusion and exclusion criteria. Screening failures were excluded from the study and were not randomized.
Groups:
- Radiofrequency (RF) Ablation Treatment: Radiofrequency (RF) ablation treatment for subjects with Paroxysmal Atrial Fibrillation (PAF) using the CARTO® 3 or CARTO® XP System, CARTO RMT, and THERMOCOOL® Catheter Family (including THERMOCOOL® SF or THERMOCOOL® SMARTTOUCH™).
- Antiarrhythmic Drug (AAD) Therapy: Antiarrhythmic Drug therapy (either rate or rhythm control): Class I or class III, or AV nodal blocking agents such as beta blockers and calcium channel blockers in accordance with 2006 atrial fibrillation management guidelines. Participants who met eligibility criteria were allowed for crossed over to RF ablation treatment (second treatment) followed by AAD therapy (first treatment).
Period: Overall Study
Arm/Group | Radiofrequency (RF) Ablation Treatment | Antiarrhythmic Drug (AAD) Therapy
Started | 128 | 127
Received Study Treatment | 102 | 123
Cross-over (AAD Therapy to RF Ablation) | 0 | 15
AAD Therapy Only | 0 | 108
Completed | 46 | 52
Not Completed | 82 | 75
Not completed — Subject discontinued | 1 | 2
Not completed — Sponsor closing the study | 51 | 50
Not completed — Subject excluded | 5 | 3
Not completed — Subject withdrew consent | 14 | 9
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 4 | 4
Not completed — Death | 5 | 4
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: The intent-to-treat population included all subjects randomized, where subjects were classified by the group to which they were randomized, regardless of the treatment received
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiofrequency (RF) Ablation Treatment | Antiarrhythmic Drug (AAD) Therapy | Total
Number analyzed (Participants) | 128 | 127 | 255
Age, Continuous [Mean (Standard Deviation); unit: Year] | 67.8 (4.83) | 67.6 (4.64) | 67.7 (4.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 74 | 148
  Male | 54 | 53 | 107
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time to Persistent Atrial Fibrillation/Atrial Tachycardia at 3 Years
Description: Persistent atrial fibrillation/atrial tachycardia (AF/AT) (excluding isthmus-dependent atrial flutter) was defined as AF/AT lasting longer than 7 consecutive days or requiring termination by cardioversion after 48 hours.
Time Frame: 3 years
Population: Intent to treat population (ITT), including all subjects randomized, where subjects were classified by the group to which they were randomized, regardless of the treatment received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radiofrequency (RF) Ablation Treatment | Antiarrhythmic Drug (AAD) Therapy
Number analyzed (Participants) | 128 | 127
Months | NA [NA to NA] — Due to insufficient number of participants with events, median time and 95% CI could not be estimated using Kaplan-Meier method. | NA [NA to NA] — Due to insufficient number of participants with events, median time and 95% CI could not be estimated using Kaplan-Meier method.
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation Treatment vs Antiarrhythmic Drug (AAD) Therapy; Test type: Superiority; p = 0.0009, Log Rank — Prior to the final analysis, study had two interim analyses. Hence alpha level is 0.0231 for primary analysis adjusted for the two interim analyses; One-sided test

2. Secondary Outcome: Time to Persistent Atrial Fibrillation/Atrial Tachycardia at 1 Year
Description: as for outcome 1
Time Frame: 1 year
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radiofrequency (RF) Ablation Treatment | Antiarrhythmic Drug (AAD) Therapy
Number analyzed (Participants) | 128 | 127
Months | NA [NA to NA] — Due to insufficient number of participants with events, median time and 95% CI could not be estimated using Kaplan-Meier method. | NA [NA to NA] — Due to insufficient number of participants with events, median time and 95% CI could not be estimated using Kaplan-Meier method.
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation Treatment vs Antiarrhythmic Drug (AAD) Therapy; Test type: Superiority; p = 0.0118, Log Rank — The alpha level is 0.025 for this secondary endpoint; One-sided test

3. Secondary Outcome: Time to Persistent Atrial Fibrillation/Atrial Tachycardia at 2 Years
Description: as for outcome 1
Time Frame: 2 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radiofrequency (RF) Ablation Treatment | Antiarrhythmic Drug (AAD) Therapy
Number analyzed (Participants) | 128 | 127
Months | NA [NA to NA] — Due to insufficient number of participants with events, median time and 95% CI could not be estimated using Kaplan-Meier method. | NA [NA to NA] — Due to insufficient number of participants with events, median time and 95% CI could not be estimated using Kaplan-Meier method.
Statistical Analysis 1: Comparison: Radiofrequency (RF) Ablation Treatment vs Antiarrhythmic Drug (AAD) Therapy; Test type: Superiority; p = 0.0041, Log Rank — The alpha level is 0.025 for this secondary endpoint; One-sided test

4. Secondary Outcome: Percentage of Participants With Persistent Atrial Fibrillation/Atrial Tachycardia at 1 Year
Description: Percentage of Participants with Persistent Atrial Fibrillation/Atrial Tachycardia at 1 year were reported. The percentage of participants was calculated using Kaplan Meier (KM) rate estimate. Persistent atrial fibrillation/atrial tachycardia (AF/AT) (excluding isthmus-dependent atrial flutter) was defined as AF/AT lasting longer than 7 consecutive days or requiring termination by cardioversion after 48 hours.
Time Frame: 1 year
Population: ITT, including all subjects randomized, where subjects were classified by the group to which they were randomized, regardless of the treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Radiofrequency (RF) Ablation Treatment | Antiarrhythmic Drug (AAD) Therapy
Number analyzed (Participants) | 128 | 127
Percentage of Participants | 1.3 [0.2 to 8.6] | 6.5 [3.2 to 13.2]

5. Secondary Outcome: Percentage of Participants With Persistent Atrial Fibrillation/Atrial Tachycardia at 2 Years
Description: Percentage of Participants with Persistent Atrial Fibrillation/Atrial Tachycardia at 2 year were reported. The percentage of participants was calculated using Kaplan Meier (KM) rate estimate. Persistent atrial fibrillation/atrial tachycardia (AF/AT) (excluding isthmus-dependent atrial flutter) was defined as AF/AT lasting longer than 7 consecutive days or requiring termination by cardioversion after 48 hours.
Time Frame: 2 Years
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Radiofrequency (RF) Ablation Treatment | Antiarrhythmic Drug (AAD) Therapy
Number analyzed (Participants) | 128 | 127
Percentage of participants | 2.4 [0.6 to 9.4] | 12.4 [7.2 to 21.0]

6. Secondary Outcome: Percentage of Participants With Persistent Atrial Fibrillation/Atrial Tachycardia at 3 Year
Description: Percentage of Participants with Persistent Atrial Fibrillation/Atrial Tachycardia at 3 year were reported. The percentage of participants was calculated using Kaplan Meier (KM) rate estimate. Persistent atrial fibrillation/atrial tachycardia (AF/AT) (excluding isthmus-dependent atrial flutter) was defined as AF/AT lasting longer than 7 consecutive days or requiring termination by cardioversion after 48 hours.
Time Frame: 3 year
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Radiofrequency (RF) Ablation Treatment | Antiarrhythmic Drug (AAD) Therapy
Number analyzed (Participants) | 128 | 127
Percentage of Participants | 2.4 [0.6 to 9.4] | 17.5 [10.7 to 27.8]

7. Secondary Outcome: Percentage of Participants With Persistent Atrial Fibrillation/Atrial Tachycardia at 3 Years by Number of Repeat Ablations
Description: Percentage of Participants with Persistent Atrial Fibrillation/Atrial Tachycardia at 3 year by number of repeat ablations were reported. The percentage of participants was calculated using Kaplan Meier (KM) rate estimate. Persistent atrial fibrillation/atrial tachycardia (AF/AT) (excluding isthmus-dependent atrial flutter) was defined as AF/AT lasting longer than 7 consecutive days or requiring termination by cardioversion after 48 hours.
Time Frame: 3 years
Population: Intent to treat population (ITT), including all subjects randomized, where subjects were classified by the group to which they were randomized, regardless of the treatment received. Endpoint applicable only to subjects randomized into the test group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Radiofrequency (RF) Ablation Treatment
Number analyzed (Participants) | 128
Percentage of participants
  Number of ablations = 0: number analyzed (Participants) | 25
  Number of ablations = 0 | 0.0 [NA to NA] — Due to insufficient number of participants with events, 95% CI could not be estimated using Kaplan-Meier method.
  Number of ablations = 1: number analyzed (Participants) | 89
  Number of ablations = 1 | 1.5 [0.2 to 10.4]
  2 or more ablations: number analyzed (Participants) | 14
  2 or more ablations | 7.7 [1.1 to 43.4]

8. Secondary Outcome: Number of Repeat Ablations
Description: Number of repeat ablations refers to the total number of ablation procedures (including initial ablation procedure). If the number of repeat ablations =1 then subject only had one ablation procedure (initial ablation procedure in test group as randomized or cross-over procedure in cross-over subjects). If the number of repeat ablations is >= 2, then subject had at least one repeat procedure.
Time Frame: 3 years
Population: Subjects in the Intent to treat population (ITT) who were randomized to RF ablation or who received any RF ablations as Cross-Over Patients randomized to AAD group. ITT population includes all subjects randomized, where subjects were classified by the group to which they were randomized, regardless of the treatment received.
Measure: Mean (Standard Deviation); unit: Event of ablation
Groups:
- Radiofrequency (RF) Ablation 2nd Treatment: Participants who were initially treated with AAD therapy (1st treatment) and then crossed over to RF ablation (2nd treatment) were evaluated. AAD therapy (either rate or rhythm control): Class I or class III, or AV nodal blocking agents such as beta blockers and calcium channel blockers in accordance with current atrial fibrillation management guidelines.
Arm/Group | Radiofrequency (RF) Ablation Treatment | Radiofrequency (RF) Ablation 2nd Treatment
Number analyzed (Participants) | 128 | 15
Event of ablation | 0.9 (0.57) | 1.1 (0.26)

9. Secondary Outcome: Number of New Antiarrhythmic Drugs
Description: Number of new antiarrhythmic drugs were administered as per investigator's discretion and 2006 AF management guidelines.
Time Frame: 3 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: AAD drug
Arm/Group | Radiofrequency (RF) Ablation Treatment | Antiarrhythmic Drug (AAD) Therapy
Number analyzed (Participants) | 128 | 127
AAD drug | 0.8 (1.05) | 1.0 (1.23)

10. Secondary Outcome: Number of Participants in Sinus Rhythm at Each Visit Throughout the Follow-up
Description: Subject in sinus rhythm: no other rhythms documented at specific visit, based on ECG, Holter and event recorder. Percentages are calculated with respect to number of subjects with data available at corresponding visit
Time Frame: 3 months, 6 months, 1 year, 2 years, 3 years
Population: Intent to treat population (ITT), including all subjects randomized, where subjects were classified by the group to which they were randomized, regardless of the treatment received. The number of participants analyzed at each visit is the number of participants with available data at the visit.
Measure: Number; unit: Participants
Arm/Group | Radiofrequency (RF) Ablation Treatment | Antiarrhythmic Drug (AAD) Therapy
Number analyzed (Participants) | 128 | 127
Participants
  3 month follow up: number analyzed (Participants) | 69 | 80
  3 month follow up | 51 | 55
  6 month follow up: number analyzed (Participants) | 62 | 60
  6 month follow up | 49 | 42
  1 year follow up: number analyzed (Participants) | 54 | 53
  1 year follow up | 41 | 35
  2 year follow up: number analyzed (Participants) | 44 | 44
  2 year follow up | 37 | 30
  3 year follow up: number analyzed (Participants) | 27 | 35
  3 year follow up | 20 | 23

11. Secondary Outcome: Number of Participants With Recurrent AF/AT at Each Visit Throughout the Follow-up
Description: Subjects with recurrent AF/AT: any AF/AT documented between previous visit up to visit analyzed at any TTM, Holter or ECG. Percentages are calculated with respect to number of subjects with data available at corresponding visit
Time Frame: 3 months, 6 months, 1 year, 2 year and 3 years
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Radiofrequency (RF) Ablation Treatment | Antiarrhythmic Drug (AAD) Therapy
Number analyzed (Participants) | 128 | 127
Participants
  3 month follow up: number analyzed (Participants) | 101 | 114
  3 month follow up | 17 | 20
  6 month follow up: number analyzed (Participants) | 96 | 110
  6 month follow up | 17 | 45
  1 year follow up: number analyzed (Participants) | 88 | 87
  1 year follow up | 20 | 38
  2 year follow up: number analyzed (Participants) | 72 | 73
  2 year follow up | 16 | 30
  3 year follow up: number analyzed (Participants) | 51 | 55
  3 year follow up | 10 | 17

ADVERSE EVENTS:
Time Frame: 3 years follow up
Description: Adverse events are summarized using the Safety population, which includes all subjects who had undergone insertion of an ablation catheter, either as RF ablation group or cross-over subjects; subjects who had started an investigator prescribed AAD in the AAD Group and did not initiate ablation therapy.
Groups:
- Antiarrhythmic Drug (AAD) Therapy Only: Antiarrhythmic Drug therapy (either rate or rhythm control): Class I or class III, or AV nodal blocking agents such as beta blockers and calcium channel blockers in accordance with 2006 atrial fibrillation management guidelines. This group includes only those subjects received AAD only.
- Antiarrhythmic Drug (AAD) Therapy - First Treatment: This group of subjects received Antiarrhythmic drug (AAD) therapy first and received RF ablation treatment later. The AEs are those occurred during the AAD treatment period.
- Radiofrequency (RF) Ablation - Second Treatment: This group of subjects received Antiarrhythmic drug (AAD) therapy first and received RF ablation treatment later. The AEs are those occurred during the RF treatment period.
Arm/Group | Radiofrequency (RF) Ablation Treatment | Antiarrhythmic Drug (AAD) Therapy Only | Antiarrhythmic Drug (AAD) Therapy - First Treatment | Radiofrequency (RF) Ablation - Second Treatment
All-Cause Mortality (participants affected / at risk) | 5/102 | 4/108 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 38/102 | 30/108 | 7/15 | 4/15
Other Adverse Events (participants affected / at risk) | 37/102 | 43/108 | 6/15 | 4/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiofrequency (RF) Ablation Treatment (N=102) | Antiarrhythmic Drug (AAD) Therapy Only (N=108) | Antiarrhythmic Drug (AAD) Therapy - First Treatment (N=15) | Radiofrequency (RF) Ablation - Second Treatment (N=15)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 8 (13) | 7 (9) | 4 (4) | 3 (4)
Atrial flutter (Cardiac disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachyarrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Prostate infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Arteriogram coronary (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nerve degeneration (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radicular syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device lead damage (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess drainage (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac ablation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiofrequency (RF) Ablation Treatment (N=102) | Antiarrhythmic Drug (AAD) Therapy Only (N=108) | Antiarrhythmic Drug (AAD) Therapy - First Treatment (N=15) | Radiofrequency (RF) Ablation - Second Treatment (N=15)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 13 (14) | 20 (22) | 2 (2) | 1 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Thyroid disorder (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram change (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heart rate irregular (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatic disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
As the study was terminated early without having met primary effectiveness or futility criteria, the study results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator (PI)/Institution and the Sponsor (or its agents) that restricts the PI's rights to discuss, present or publish trial results after the trial is completed. Please contact Biosense Webster, Inc. for additional information.

DOCUMENTS (2):
  • Study Protocol (2013-04-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT01570361/Prot_001.pdf
  • Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT01570361/SAP_000.pdf